CLINICAL TRIAL: NCT03894176
Title: Association of Plasma Pentraxin 3 Concentration With Angiographic and Clinical Outcomes in STEMI Treated by Primary Angioplasty
Brief Title: Association of Plasma PTX3 Concentration and Outcomes of STEMI
Status: Completed | Type: Observational
Sponsor: Indonesian Cardiovascular Research Center (Other)
Responsible Party: Principal Investigator, Surya Dharma, Primary Investigator, Indonesian Cardiovascular Research Center
Other Study IDs: IndonesianCRC
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: STEMI; Coronary; Ischemic
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PTX3 concentration: First quartile, second quartile, third quartile and fourth quartile of PTX3 in ng/mL
  Interventions: Other: Plasma PTX3 concentration

INTERVENTIONS:
Other: Plasma PTX3 concentration — Long pentraxin 3, thrombus burden, final TIMI flow, ST segment resolution, STEMI, primary PCI
  Other Names: PTX3

SUMMARY:
335 of patients with STEMI treated by primary PCI were assayed for PTX3 measurement by ELISA method. The angiographic and clinical outcomes were evaluated according to the PTX3 concentration.

DETAILED DESCRIPTION:
335 of patients with STEMI treated by primary PCI were assayed for PTX3 measurement by ELISA method using human PTX3 kit. Blood was drawn at the emergency department before primary PCI. The angiographic and clinical outcomes were evaluated and analyzed according to the PTX3 concentration. The angiographic outcome were thrombus grade on initial angiogram and final TIMI flow. The clinical outcome were ECG resolution after primary PCI and all-cause death at 30 days. The plasma PTX3 concentration was then compared based on the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute STEMI with symptom onset <12 h undergoing primary PCI

Exclusion Criteria:

* Acute STEMI patients who received fibrinolytic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with STEMI with symptom onset <12 h who admiited to the emergency department and planned for primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
The proportion of thrombus grade 4&5 and final TIMI flow <3 | Intraprocedure
  PTX3 concentration was compared based on the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Indonesian Cardiovascular Research Center, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No